CLINICAL TRIAL: NCT07337200
Title: The Effectiveness of Daily Three Good Thing Intervention on Gratitude and Psychological Well-being Among Indonesian Nursing Students: Solomon Four-Group Design
Brief Title: The Effectiveness of Three Good Things on Gratitude and Psychological Well-being Among Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Yudisa Diaz Lutfi Sandi, Principal Investigator, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25.11.02
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Nursing Student; Gratitude; Psychological Well-being
Keywords: Three Good Things; Gratitude; Psychological well-being; Daily intervention; Nursing students; Solomon Four Group Design; Positive psychology
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study used the Solomon Four Group Design, which involved four separate groups to test the effects of the intervention while simultaneously controlling and measuring the interaction effects of the pre-test (testing effect).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Pre-test, 3GT, post-test) (Experimental): This group received measurements of the dependent variables (Gratitude and Psychological Well-being) through a pre-test, followed by a Three Good Things (3GT) intervention for 7 days, and ended with the same measurements for the post-test.
  Interventions: Behavioral: Three Good Things
- Group 2 (pre-test and post-test) (No Intervention): This group received measurements of dependent variables (Gratitude and Psychological Wellbeing) through a pre-test, did not receive the 3GT intervention, and ended with the same measurements. This group aimed to measure the natural effects of the passage of time and the potential influence of the pre-test itself without any intervention.
- Group 3 (3GT and post-test) (Experimental): This group does not receive a pre-test to eliminate testing bias, but receives the Three Good Things (3GT) Intervention for 7 days, and ends with only dependent variable measurements (post-test). This group tests the effectiveness of the intervention without the interaction effect of the pre-test.
  Interventions: Behavioral: Three Good Things
- Group 4 (Post Test only) (No Intervention): This group did not receive a pre-test or the 3GT Intervention. They only received a measurement of the dependent variable through a post-test at the end of the study period. This group served as the baseline measurement to isolate the pure effect of the intervention.

INTERVENTIONS:
Behavioral: Three Good Things — The Three Good Things intervention was self-administered daily for seven days. Participants are required to record three positive things that happened that day and add a brief summary of the reasons behind these events using a Google form prepared by the researchers.
  Arms: Group 1 (Pre-test, 3GT, post-test); Group 3 (3GT and post-test)

SUMMARY:
The goal of this clinical trial is to learn if the daily Three Good Thing intervention can prevent negative mental health outcomes like stress and burnou, and promote Gratitude and Psychological Wellbeing in undergraduate Nursing Students.

The main questions it aims to answer are:

Does the daily Three Good Things intervention effective in promoting gratitude and psychological wellbeing among nursing students?

Researchers will compare four different arms from Solomon Four Group Design to see if the increase in Gratitude and Psychological Wellbeing scores is significantly greater in the groups that received the 3GT intervention.

Participants will be randomly assigned to one of the four groups, and those in the intervention groups will:

1. Complete a pre-test questionnaire (for some groups) on their current level of Gratitude and Psychological Wellbeing.
2. Perform the Three Good Things (3GT) intervention by writing down three positive things that happened each day for 7 consecutive days.
3. Complete a post-test questionnaire to measure the final level of Gratitude and Psychological Wellbeing.

DETAILED DESCRIPTION:
Research Design: Experimental research using the Solomon Four Group Design approach. This design is used to measure the effectiveness of interventions while specifically controlling and analyzing the potential interaction effects between pre-tests and interventions (testing effect). Population & Sample: The population of this study consisted of all first- and second-year students of the D-III Nursing Study Program at Subang State Polytechnic, totaling 277 people. Intervention Duration: The Three Good Things intervention was carried out for 7 consecutive days.

Independent Variable: Three Good Things Daily Intervention.

Dependent Variables:

1. Gratitude: Measured using the Indonesian adaptation of the Gratitude Questionnaire containing 11 items.
2. Psychological Wellbeing: Measured using the Indonesian adaptation of Ryff's Psychological Wellbeing Scale questionnaire containing 18 items.

ELIGIBILITY:
Inclusion Criteria:

* Active first- and second-year students in the D-III Nursing Program at Subang State Polytechnic.
* Willing to participate in the study by signing an informed consent form.
* Able to use Google Forms online for the intervention.

Exclusion Criteria:

* Students who are on academic leave.
* Students who did not complete the daily intervention until the end in groups 1 and 3.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
The Change in Psychological Well-Being | 7 days (Measured immediately after completion of the one-week daily intervention)
  Measurement of changes in psychological well-being scores from pre-test to post-test in participants using the 18-item Indonesian adaptation of the Ryff Psychological Well-Being Scale. These changes will compare the effectiveness of the Three Good Things (3GT) intervention with the control group. Psychological well-being here refers to six dimensions : self-acceptance, positive relationships with others, autonomy, mastery of the environment, life purpose, and personal growth. The total score ranges from 18 to 72 using a 1-4 Likert scale (strongly disagree-strongly agree), where a higher score indicates a higher level of psychological well-being. Reverse scoring is used for favorable items 4, 5, 6, 7, 10, 14, 15, and 16.
The Change in Gratitude Levels | 7 days (Measured immediately after completion of the daily intervention for one week)
  Measurement of changes in gratitude scores from pre-test to post-test in participants using the 11-item Indonesian adaptation of the Gratitude Questionnaire. These changes will assess the ability of the Three Good Things (3GT) intervention to increase participants' tendency to feel and express gratitude in their daily lives using two dimensions : Appreciation for ongoing life experiences and Appreciation for individuals involved in one's life. The total score ranges from 11 to 77 using a 1-7 Likert scale (strongly disagree-strongly agree), where a higher score indicates a higher level of gratitude. Reverse scoring applies to unfavorable item number 3.

CONTACTS AND LOCATIONS:
Overall Officials: Yudisa Diaz Lutfi Sandi RN, MSN, RN., PhD, Principal Investigator — School of Health Science, Politeknik Negeri Subang
Locations (1):
- Subang State Polytechnic, Subang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared to maintain participant confidentiality and to comply with the ethical guidelines. Furthermore, the study protocol and informed consent process do not include provisions for sharing participant data with external parties.

REFERENCES:
- [Background] Zhan D, Xu L, Ouyang Y, Sawatzky R, Wong H. Methods for dealing with unequal cluster sizes in cluster randomized trials: A scoping review. PLoS One. 2021 Jul 29;16(7):e0255389. doi: 10.1371/journal.pone.0255389. eCollection 2021. PMID 34324593
- [Background] Yosep I, Hikmat R, Mardhiyah A, Zamroni AH, Pranata Y, Saputra RL. Nursing interventions to reduce mental health problems in nursing students: a scoping review. BMC Nurs. 2025 Jul 1;24(1):780. doi: 10.1186/s12912-025-03329-w. PMID 40598211
- [Background] Xiong, Y., & Higgins, M. J. (2020). The Benefits of Probability-Proportional-to-Size Sampling in Cluster-Randomized Experiments (No. arXiv:2002.08009). arXiv. https://doi.org/10.48550/arXiv.2002.08009
- [Background] Xie H, Kang B. Mental Health of Nursing Students: A Bibliometric Review Based on CiteSpace Visual Analysis. J Nurs Manag. 2025 Mar 12;2025:2169094. doi: 10.1155/jonm/2169094. eCollection 2025. PMID 40223903
- [Background] World Health Organization. (2025). Mental Health of Adolescents. https://www.who.int/news-room/fact-sheets/detail/adolescent-mental-health
- [Background] Willenberg L, Wulan N, Medise BE, Devaera Y, Riyanti A, Ansariadi A, Wiguna T, Kaligis F, Fisher J, Luchters S, Jameel A, Sawyer SM, Tran T, Kennedy E, Patton GC, Wiweko B, Azzopardi PS. Understanding mental health and its determinants from the perspective of adolescents: A qualitative study across diverse social settings in Indonesia. Asian J Psychiatr. 2020 Aug;52:102148. doi: 10.1016/j.ajp.2020.102148. Epub 2020 May 6. PMID 32450491
- [Background] Sucitayasa, I. M. (2025). Hubungan Dukungan Sosial Dengan Tingkat Stres Mahasiswa Tingkat Satu Program Studi Sarjana Keperawatan Dan Pendidikan Profesi Ners Fakultas Kedokteran Universitas Udayana. Community of Publishing in Nursing, 13(1), 102-109.
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Safrin. (2020). Pendekatan Eksperimental dalam Penelitian Komunikasi. Talenta Conference Series: Local Wisdom, Social, and Arts (LWSA), 3(1). https://doi.org/10.32734/lwsa.v3i1.810
- [Background] Rippstein-Leuenberger K, Mauthner O, Bryan Sexton J, Schwendimann R. A qualitative analysis of the Three Good Things intervention in healthcare workers. BMJ Open. 2017 Jun 13;7(5):e015826. doi: 10.1136/bmjopen-2017-015826. PMID 28611090
- [Background] Rahmi, E. F., & Appulembang, Y. A. (2024). Konseling Kelompok Untuk Menurunkan Stress Akademik Mahasiswa Tingkat Akhir S. PUSAKO : Jurnal Pengabdian Psikologi, 2(2), 39-48. https://doi.org/10.24036/pusako.v2i2.55
- [Background] Radez J, Reardon T, Creswell C, Lawrence PJ, Evdoka-Burton G, Waite P. Why do children and adolescents (not) seek and access professional help for their mental health problems? A systematic review of quantitative and qualitative studies. Eur Child Adolesc Psychiatry. 2021 Feb;30(2):183-211. doi: 10.1007/s00787-019-01469-4. Epub 2020 Jan 21. PMID 31965309
- [Background] Pusat Kesehatan Reproduksi UGM. (2021). Indonesia-National Adolescent Mental Health (I-NAMHS). https://pkr.fk.ugm.ac.id/penelitian/indonesia-national-adolescent-mental-health/#:~:text=Penelitian%20Indonesia%2DNational%20Adolescent%20Mental%20Survey%20(I%2DNAMHS),prevalensi%20penyakit%20mental%20pada%20remaja.
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629
- [Background] Mat, N., Abdullah, N. A., Abu Hassan, N., & Juhdi, N. H. (2020). Pengaruh Nilai Kerja Terhadap Tingkah Laku Kerja Inovatif dan Kesejahteraan Psikologi: Modal Psikologi Sebagai Pengantara (the Influence of Work Values on Innovative Work Behaviour and Psychological Well-Being: The Psychological Capital as a Mediator). International Journal of Management Studies, 27. https://doi.org/10.32890/ijms.27.1.2020.7674
- [Background] Lockertsen O, Lovhaug L, Davik NK, Bolgen BR, Faerden A, Skarstein S. Second-year undergraduate nursing students' experiences with clinical simulation training in mental health clinical practice: A focus group study. Nurse Educ Pract. 2023 Jan;66:103534. doi: 10.1016/j.nepr.2022.103534. Epub 2022 Dec 12. PMID 36563598
- [Background] Lee N, Kim Y. A Meta-Analysis on the Effectiveness of Gratitude Promotion Programs for South Korean College Students. Behav Sci (Basel). 2024 Mar 15;14(3):240. doi: 10.3390/bs14030240. PMID 38540543
- [Background] Humaidah, A., & Mulyono, R. (2025). Adaptasi Psychological Well-Being Short Scale pada Mahasiswa. 7(1).
- [Background] Hemarajarajeswari, J., & Gupta, P. K. (2021). Gratitude, Psychological Well-Being and Happiness Among College Students: A Correlational Study. The International Journal of Indian Psychology, 9(1). https://doi.org/10.25215/0901.053
- [Background] Hamshire C, Jack K, Forsyth R, Langan AM, Harris WE. The wicked problem of healthcare student attrition. Nurs Inq. 2019 Jul;26(3):e12294. doi: 10.1111/nin.12294. Epub 2019 May 6. PMID 31056831
- [Background] Grimaldy, D. V., & Haryanto, H. C. (2020). Adaptation of Gratitude Questionnaire-6 (GQ-6) in Indonesian Context. Jurnal Psikologi, 47(1), 18. https://doi.org/10.22146/jpsi.39608
- [Background] Gold KJ, Dobson ML, Sen A. "Three Good Things" Digital Intervention Among Health Care Workers: A Randomized Controlled Trial. Ann Fam Med. 2023 May-Jun;21(3):220-226. doi: 10.1370/afm.2963. PMID 37217328
- [Background] Ghania, S., & Prihatsanti, U. (2025). Faktpr-Faktor Yang Mempengaruhi Stres Akademik Pada Mahasiswa Di Indonesia: Studi Literatur. Jurnal Empati, 14(03), 265-273.
- [Background] Garcia D, Kazemitabar M, Asgarabad MH. The 18-item Swedish version of Ryff's psychological wellbeing scale: psychometric properties based on classical test theory and item response theory. Front Psychol. 2023 Oct 3;14:1208300. doi: 10.3389/fpsyg.2023.1208300. eCollection 2023. Erratum In: Front Psychol. 2023 Nov 03;14:1324006. doi: 10.3389/fpsyg.2023.1324006. PMID 37854148
- [Background] Frey, B. B. (2018). The SAGE Encyclopedia of Educational Research, Measurement, and Evaluation. SAGE Publications, Inc. https://doi.org/10.4135/9781506326139
- [Background] Erskine HE, Maravilla JC, Wado YD, Wahdi AE, Loi VM, Fine SL, Li M, Ramaiya A, Wekesah FM, Odunga SA, Njeri A, Setyawan A, Astrini YP, Rachmawati R, Hoa DTK, Wallis K, McGrath C, Shadid J, Enright ME, Blondell SJ, Lawrence D, Fisher PW, Whiteford HA, Vinh ND, Wilopo SA, Kabiru CW, Blum RW, Scott JG. Prevalence of adolescent mental disorders in Kenya, Indonesia, and Viet Nam measured by the National Adolescent Mental Health Surveys (NAMHS): a multi-national cross-sectional study. Lancet. 2024 Apr 27;403(10437):1671-1680. doi: 10.1016/S0140-6736(23)02641-7. Epub 2024 Apr 5. PMID 38588689
- [Background] El Karkri, M., Quesada, A., & Romero-Ariza, M. (2025). Methodological Aspects of the Solomon Four-Group Design: Detecting Pre-Test Sensitisation and Analysing Qualitative and Quantitative Variables in Education Research. Review of Education, 13(1), e70050. https://doi.org/10.1002/rev3.70050
- [Background] Efstathiou M, Kakaidi V, Tsitsas G, Mantzoukas S, Gouva M, Dragioti E. The prevalence of mental health issues among nursing students: An umbrella review synthesis of meta-analytic evidence. Int J Nurs Stud. 2025 Mar;163:104993. doi: 10.1016/j.ijnurstu.2025.104993. Epub 2025 Jan 7. PMID 39809132
- [Background] Dutta, U., & Teotia, A. (2022). Gratitude, Life Satisfaction And Forgiveness Among Acid Attack Victims: Rehabilitation Through Three Good Things Intervention. Online Journal of Health and Allied Sciences, 21(3). https://www.ojhas.org/issue83/2022-3-5.html
- [Background] Donmez AA, Alici NK, Kapucu S, Elcin M. The effect of laughter yoga applied before simulation training on state anxiety, perceived stress levels, self-confidence and satisfaction in undergraduate nursing students: A pragmatic randomized controlled trial. Nurse Educ Pract. 2023 Jul;70:103636. doi: 10.1016/j.nepr.2023.103636. Epub 2023 Apr 12. PMID 37100026
- [Background] Cohen, J. (2009). Statistical Power Analysis for the Behavioral Sciences (2. ed., reprint). Psychology Press.
- [Background] Canzan F, Saiani L, Mezzalira E, Allegrini E, Caliaro A, Ambrosi E. Why do nursing students leave bachelor program? Findings from a qualitative descriptive study. BMC Nurs. 2022 Mar 29;21(1):71. doi: 10.1186/s12912-022-00851-z. PMID 35351118
- [Background] Bartlett ML, Taylor H, Nelson JD. Comparison of Mental Health Characteristics and Stress Between Baccalaureate Nursing Students and Non-Nursing Students. J Nurs Educ. 2016 Feb;55(2):87-90. doi: 10.3928/01484834-20160114-05. PMID 26814818
- [Background] Badan Pusat Statistik Provinsi Jawa Barat. (2024). Jumlah Penduduk Disabilitas Jawa Barat Menurut Kabupaten/Kota (Jiwa), 2022. https://jabar.bps.go.id/id/statistics-table/2/ODk4IzI=/jumlah-penduduk-disabilitas-jawa-barat-menurut-kabupaten-kota.html
- [Background] Aloufi MA, Jarden RJ, Gerdtz MF, Kapp S. Reducing stress, anxiety and depression in undergraduate nursing students: Systematic review. Nurse Educ Today. 2021 Jul;102:104877. doi: 10.1016/j.nedt.2021.104877. Epub 2021 Mar 18. PMID 33905898
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- See also: Consort 2010 Statement: Extension to Cluster Randomised Trials — https://doi.org/10.1136/bmj.e5661
- See also: Reducing Stress, Anxiety and Depression in Undergraduate Nursing Students: Systematic Review — https://doi.org/10.1016/j.nedt.2021.104877
- See also: Why Do Nursing Students Leave Bachelor Program? Findings from a Qualitative Descriptive Study — https://doi.org/10.1186/s12912-022-00851-z
- See also: The Effect of Laughter Yoga Applied Before Simulation Training on State Anxiety, Perceived Stress Levels, Self-Confidence and Satisfaction in Undergraduate Nursing Students: A Pragmatic Randomized Controlled Trial — https://doi.org/10.1016/j.nepr.2023.103636
- See also: Gratitude, Life Satisfaction And Forgiveness Among Acid Attack Victims: Rehabilitation Through Three Good Things Intervention — https://www.ojhas.org/issue83/2022-3-5.html
- See also: The Prevalence of Mental Health Issues Among Nursing Students: An Umbrella Review Synthesis of Meta-Analytic Evidence — https://doi.org/10.1016/j.ijnurstu.2025.104993
- See also: Prevalence of Adolescent Mental Disorders in Kenya, Indonesia, and Viet Nam Measured by the National Adolescent Mental Health Surveys (NAMHS): A Multi-National Cross-Sectional Study — https://doi.org/10.1016/S0140-6736(23)02641-7
- See also: The SAGE Encyclopedia of Educational Research, Measurement, and Evaluation — https://doi.org/10.4135/9781506326139
- See also: The 18-Item Swedish Version of Ryff's Psychological Wellbeing Scale: Psychometric Properties Based on Classical Test Theory and Item Response Theory — https://doi.org/10.3389/fpsyg.2023.1208300
- See also: Factors Affecting Academic Stress in Students in Indonesia: A Literature Study — https://ejournal3.undip.ac.id/index.php/empati/article/view/50074
- See also: Second-Year Undergraduate Nursing Students' Experiences with Clinical Simulation Training in Mental Health Clinical Practice: A Focus Group Study — https://doi.org/10.1016/j.nepr.2022.103534
- See also: the Influence of Work Values on Innovative Work Behaviour and Psychological Well-Being: The Psychological Capital as a Mediator — https://doi.org/10.32890/ijms.27.1.2020.7674
- See also: Indonesia-National Adolescent Mental Health (I-NAMHS) — https://pkr.fk.ugm.ac.id/penelitian/indonesia-national-adolescent-mental-health/#:~:text=Penelitian%20Indonesia%2DNational%20Adolescent%20Mental%20Survey%20(I%2DNAMHS),prevalensi%20penyakit%20mental%20pada%20remaja.
- See also: Why Do Children and Adolescents (not) Seek and Access Professional Help for Their Mental Health Problems? A Systematic Review of Quantitative and Qualitative Studies — https://doi.org/10.1007/s00787-019-01469-4
- See also: Group Counseling to Reduce Academic Stress in Final Year Students — https://doi.org/10.24036/pusako.v2i2.55
- See also: A Qualitative Analysis of the Three Good Things Intervention in Healthcare Workers — https://doi.org/10.1136/bmjopen-2017-015826
- See also: Experimental Approaches in Communication Research — https://doi.org/10.32734/lwsa.v3i1.810
- See also: Understanding Mental Health and Its Determinants from the Perspective of Adolescents: A Qualitative Study Across Diverse Social Settings in Indonesia — https://doi.org/10.1016/j.ajp.2020.102148
- See also: Mental Health of Adolescents — https://www.who.int/news-room/fact-sheets/detail/adolescent-mental-health
- See also: The Benefits of Probability-Proportional-to-Size Sampling in Cluster-Randomized Experiments — https://doi.org/10.48550/arXiv.2002.08009
- See also: Nursing Interventions to Reduce Mental Health Problems in Nursing Students: A Scoping Review — https://doi.org/10.1186/s12912-025-03329-w
- See also: Methods for Dealing with Unequal Cluster Sizes in Cluster Randomized Trials: A Scoping Review — https://doi.org/10.1371/journal.pone.0255389